CLINICAL TRIAL: NCT01520688
Title: A Randomized, Cross Over Study Evaluating the Effect of Flovent Discus 100 mcg BID vs QVAR 80 mcg BID vs Pulmicort Flexhaler 180 mcg BID on Short Term Growth in Pediatric Subjects With Asthma
Brief Title: Effect of Flovent Discus vs QVAR vs Pulmicort Flexhaler on Short Term Growth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Deborah Gentile, Principal Investigator, West Penn Allegheny Health System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC#5255
Record Dates: First submitted 2012-01-24; First posted 2012-01-30 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: Mild persistent or mild intermittent asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Budesonide; Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 Treatment Sequence, FPQ (Experimental): Period 2 Flovent Diskus Period 4 Pulmicort Flexhaler Period 6 QVAR
  Interventions: Drug: Fluticasone, Budesonide, Beclomethasone
- 2 Treatment Sequence, FQP (Experimental): Period 2 Flovent Diskus Period 4 QVAR Period 6 Pulmicort
  Interventions: Drug: Fluticasone, Beclomethasone, Budesonide
- 3 Treatment Sequence, PFQ (Experimental): Period 2 Pulmicort Period 4 Flovent Period 6 QVAR
  Interventions: Drug: Budesonide, Fluticasone, Beclomethasone
- 4-Treatment Sequence, PQF (Experimental): Period 2 Pulmicort Period 4 QVAR Period 6 Flovent
  Interventions: Drug: Budesonide, Beclomethasone, Fluticasone
- 5 Treatment Sequence, QFP (Experimental): Period 2 QVAR Period 4 Flovent Period 6 Pulmicort
  Interventions: Drug: Beclomethasone, Fluticasone, Budesonide
- 6 Treatment Sequence, QPF (Experimental): Period 2 QVAR Period 4 Pulmicort Period 6 Flovent
  Interventions: Drug: Beclomethasone, Budesonide, Fluticasone

INTERVENTIONS:
Drug: Fluticasone, Budesonide, Beclomethasone — Fluticasone 100 mcg bid Budesonide 180 mcg bid Beclomethasone 80 mcg bid
  Other Names: Flovent Diskus; Pulmicort Flexhaler; QVAR
  Arms: 1 Treatment Sequence, FPQ
Drug: Fluticasone, Beclomethasone, Budesonide — Fluticasone 100mcg BID Beclomethasone 80 mcg BID Budesonide 180 mcg BID
  Other Names: Flovent Diskus; Pulmicort Flexhaler; QVAR
  Arms: 2 Treatment Sequence, FQP
Drug: Budesonide, Fluticasone, Beclomethasone — Budesonide180 mcg BID Fluticasone 100 mcg Beclomethasone 80 mcg BID
  Other Names: Pulmicort Flexhaler; Flovent Diskus; QVAR
  Arms: 3 Treatment Sequence, PFQ
Drug: Budesonide, Beclomethasone, Fluticasone — Budesonide 180 mcg BID Beclomethasone 80mcg BID Fluticasone 100mcg BID
  Other Names: Pulmicort Flexhaler; QVAR; Flovent Diskus
  Arms: 4-Treatment Sequence, PQF
Drug: Beclomethasone, Fluticasone, Budesonide — Beclomethasone 80 mcg BID Fluticasone 100mcg BID Budesonide 180 mcg BID
  Other Names: QVAR; Flovent Diskus; Pulmicort Flexhaler
  Arms: 5 Treatment Sequence, QFP
Drug: Beclomethasone, Budesonide, Fluticasone — Beclomethasone 80mcg BID Budesonide 180 mcg BID Fluticasone 100mcg BID
  Other Names: QVAR; Pulmicort Flexhaler; flovent Diskus
  Arms: 6 Treatment Sequence, QPF

SUMMARY:
Children with mild persistent asthma that have asthma symptoms once or twice a week and use a daily controller, while children with mild intermittent asthma rarely have asthma symptoms and do not use a daily controller. Inhaled corticosteroids are the standard treatment for mild peristent asthma. The purpose of this study is to measure children rate of growth while on different inhaled corticosteroids.

DETAILED DESCRIPTION:
A randomized, cross over study evaluating the effect of Flovent Discus 100 mcg BID vs QVAR 80 mcg BID vs Pulmicort Flexhaler 180 mcg BID on short term growth in pediatric subjects with asthma.

Objectives:

1. The primary objective of this study is to compare the effect of Flovent Diskus 100 mcg BID versus Pulmicort Flexhaler 180 mcg BID on short-term lower leg growth velocity as measured by knemometry in pediatric subjects with mild asthma.
2. The secondary objective of this study is to compare the effect of Flovent Diskus 100 mcg BID versus QVAR 80 mcg BID on short-term lower leg growth velocity as measured by knemometry in pediatric subjects with mild asthma.

Aims:

1. The primary aim is to show that there is a growth suppressive effect of Pulmicort Flexhaler 180 mcg BID versus Flovent Diskus 100 mcg BID in children with mild asthma.
2. The secondary aim to show that there is a growth suppressive effect of QVAR 80 mcg BID versus Flovent Diskus 100 mcg BID in children with mild asthma.

Hypotheses:

1. The primary hypothesis is that treatment with Pulmicort Flexhaler 180mcg BID as compared to Flovent Diskus 100 mcg BID has a growth suppressive effect on lower leg length as assessed by knemometry in pediatric subjects with mild asthma.
2. The secondary hypothesis is that treatment with QVAR 80 mcg BID as compared to Flovent Diskus 100 mcg BID has a growth suppressive effect on lower leg length as assessed by knemometry in pediatric subjects with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will include females (6 to 9 years of age) and males (6 to 11 years of age).
2. All subjects must have a history of physician diagnosed mild intermittent or mild persistent asthma as documented by PCP medical record or detailed history by study investigator.
3. All subjects must have a height within normal limits (5th to 95th percentile) and no history of abnormal growth as assessed by medical history.
4. All subjects must be pre-pubertal (Tanner Stage 1 Sexual Maturity) as assessed by physical examination.
5. Subjects may be on current treatment with montelukast as this drug does not affect growth. If a subject is on montelukast at screening/baseline, they will remain on a stable dose throughout the study.
6. Subjects must be willing to comply with study requirements.

Exclusion Criteria:

1. Subjects will be excluded if they have asthma greater than mild persistent severity as defined by NHLBI guidelines.
2. Subjects will be excluded if they used any systemic or nasal steroids within the past 60 days.
3. Subjects will be excluded if they had more than one burst of systemic steroids within the past year.
4. Subjects will be excluded if their baseline FEV1 is < 80% predicted.
5. Subjects will be excluded if they have any other serious systemic disease other than asthma.
6. Subjects will be excluded if they have taken any medication known to affect growth i.e. ADHD medications within the past 60 days
7. Subjects will be excluded if they have a history of allergy to any of the study medications, milk protein or lactose.
8. Subjects will be excluded if they have active chickenpox or measles or recent exposure to chickenpox or measles.
9. Subjects will be excluded if they have any history of tuberculosis of the respiratory tract.
10. Subjects will be excluded if they have any active fungal, bacterial, viral or parasitic infections.
11. Subjects will be excluded if they have any history of herpes simplex infection of the eye.
12. Subjects will be excluded if they have taken any immunosuppressive drugs within the past 2 months.
13. Subjects will be excluded if they have any history of Churg-Strauss syndrome or other eosinophilic disorders.
14. Subjects will be excluded if an investigator deems they have any mental or development health issues, such as autism, moderate to severe mental retardation or severe ADHD,that interferes with their ability to complete the knemometry measurements.
15. Subjects will be excluded if an investigator deems they have any physical issues, such as inability to sit independently or amputation of lower leg, that interferes with their ability to complete the knemometry measurements.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Gentile, MD, Principal Investigator — Allegheny Singer Research Institute/Allegheny General Hospital
Locations (2):
- United States (2):
  - Pediatric Alliance-Greentree Division, Green Tree, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled But Not Randomized.: These subjects were consented but not randomized.
Period: Overall Study
Arm/Group | 1 Treatment Sequence, FPQ | 2 Treatment Sequence, FQP | 3 Treatment Sequence, PFQ | 4-Treatment Sequence, PQF | 5 Treatment Sequence, QFP | 6 Treatment Sequence, QPF | Enrolled But Not Randomized.
Started | 4 | 4 | 4 | 5 | 5 | 5 | 5
Completed | 4 | 2 | 4 | 4 | 4 | 5 | 0
Not Completed | 0 | 2 | 0 | 1 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Short-term Lower Leg Growth During Treatment With Flovent Diskus 100 mcg BID or Pulmicort Flexhaler 180 mcg BID.
Description: Short-term lower leg growth as assessed by knemometry in pediatric subjects with mild asthma treated with Flovent Discus 100 mcg BID or Pulmicort Flexhaler 180 mcg BID.
Time Frame: 1 yr
Measure: Mean (95% Confidence Interval); unit: mm/wk
Arm/Group | Flovent Discus 100 mcg BID | Pulmicort Flexhaler 180 mcg BID
Number analyzed (Participants) | 27 | 27
mm/wk | 0.37 [0.21 to 0.53] | 0.21 [0.05 to 0.37]

2. Secondary Outcome: Short-term Lower Leg Growth During Treatment With Flovent Discus 100 mcg BID or QVAR 80 mcg BID.
Description: Short-term lower leg growth as assessed by knemometry in pediatric subjects with mild asthma during treatment with Flovent Discus 100 mcg BID or QVAR 80 mcg BID.
Time Frame: 1 yr
Measure: Mean (95% Confidence Interval); unit: mm/wk
Arm/Group | Flovent Discus 100 mcg BID | QVAR 80 mcg BID
Number analyzed (Participants) | 27 | 27
mm/wk | 0.37 [0.21 to 0.53] | 0.38 [0.22 to 0.54]

ADVERSE EVENTS:
Arm/Group | Flovent Discus 100 mcg BID | Pulmicort Flexhaler 180 mcg BID | QVAR 80 mcg BID
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 7/27 | 6/27 | 7/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flovent Discus 100 mcg BID (N=27) | Pulmicort Flexhaler 180 mcg BID (N=27) | QVAR 80 mcg BID (N=27)
Colds/viral illnesses (General disorders) | 7 | 6 | 7
Headaches (General disorders) | 2 | 3 | 3
Respiratory infections (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Worsening allergies (Immune system disorders) | 1 | 0 | 1
Bodily injuries (General disorders) | 1 | 1 | 0
Asthma exacerbation (Immune system disorders) | 1 | 0 | 0
Ear infection (Ear and labyrinth disorders) | 0 | 0 | 1
Sinus infection (General disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No